CLINICAL TRIAL: NCT06761820
Title: Evaluation the Effect of Glycemic Control on Cardiac Function in Patients with Type 2 Diabetes Mellitus
Brief Title: Effect the Glycemic Control on Cardiac Function
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ramez Gamal Shawky, Doctor, Assiut University
Other Study IDs: Glycemic control and EF
Record Dates: First submitted 2024-12-24; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Cardiac Function; Glycemic Control
MeSH Terms: interventions — Echocardiography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Echocardiogram — Echo : for evaluation anatomical and functional alteration LV and diastolic dysfunction and myocardial reserve measure by LVEF by M-mode before the study and follow up echo assessment 3 months after glycemic control

SUMMARY:
Evaluation of the effect of the Glycemic control on cardiac function in patients with type 2 diabetes mellitus

DETAILED DESCRIPTION:
Type 2 Diabetes Mellitus (T2DM) is one of the most common metabolic disorders worldwide and its development is primarily caused by a combination of two main factors: defective insulin secretion by pancreatic β-cells and the inability of insulin-sensitive tissues to respond to insulin diabetes mellitus is a chronic, metabolic disease characterized by elevated levels of blood glucose, which leads over time to damage to the heart,vasculature, eyes, kidneys and nerves.

Over 90% of diabetes mellitus cases are T2DM, a conditionmarked by deficient insulin secretion by pancreatic islet β-cells, tissue insulin resistance (IR) and aninadequate compensatory insulin secretory response . Progression of the disease makes insulinsecretion unable to maintain glucose homeostasis, producing hyperglycaemia.

T2DM is a multisystem disease with a strong correlation with CVD development T2DM leads to a two- to four-fold increase in the mortality rate of adults from heart disease and is associated with both micro- and macro-vascular complications, the latter consisting of accelerated atherosclerosis leading to severe peripheral vascular disease, premature coronary artery disease (CAD) . These factors lead to T2DM being considered a significant risk factor for CVD ]. These include the role of IR in atherosclerosis, vascular function, oxidative stress, hypertension, macrophage accumulation and inflammation Factors implicated in cardiovascular risk outcomes from T2DM and the interactions between them. T2DM derived hyperglycemia, hyperinsulinemia and IR causes endothelial dysfunction, diabetic dyslipidemia and inflammation leading to atherosclerosis leading to CVD.

In addition, it is well documented that type 2 DM is associated with enhancement of platelet and hemostatic activities

Clinical trials have shown that intensive glucose control reduces the risk for microvascular complications among patients with type 2 diabetes, but its effect on CVD, including coronary heart disease (CHD), and peripheral arterial disease, is uncertain . Early data from the UKPDS (United Kingdom Prospective Diabetes Study) 34 suggested a protective effect of improved glucose control on CVD, CVD deaths, and all-causes mortality

Poor glycemic control and insulin resistance are associated with deterioration of heart failure and LV dysfunction . However, available data suggest no difference in the risk of worsening heart failure between subjecting patients to intensive glycemic control and standard treatment arms . The relationship between glycated hemoglobin (Hba1c) and LVEF remains unclear

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetic patients with heart diseases

Exclusion Criteria:

* patients with type 1 diabetes mellitus
* gestational DM
* CKD patients requiring haemodialysis
* Immune system disorder

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Cardiology and diabetes outpatients clinics, internal medicine. Assiut University hospital.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
functional alteration of left ventricel | 3 months
  Echocardiography for evaluation anatomical (chamber demision by M - mode) and functional alteration LV and diastolic dysfunction and myocardial reserve measure by LVEF before the study and follow up echo assessment 3 month after glycemic control.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Hossam Hassan, Professor, Study Chair — Assiut University; Hanaa Mohamed Riad, Doctor (lecture), Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided